CLINICAL TRIAL: NCT03259737
Title: An Observational Study of Stroke Patients With Focus on Examinations and Therapeutic Improvement the First 72 Hours.
Brief Title: An Observational Study of Stroke Patients.
Acronym: SPET-72
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ellen Bøhmer (Other)
Responsible Party: Sponsor-Investigator, Ellen Bøhmer, PHD cand med, Sykehuset Innlandet HF
Organization: Sykehuset Innlandet HF (Other)
Other Study IDs: REK2015/358
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Quality of Care; Cerebrovascular Disorders; Hyperglycemia; Hypertension; Troponin
MeSH Terms: conditions — Cerebrovascular Disorders; Hyperglycemia; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The intention is to study presumed changes in daily practice, probably due to New Guidelines concerning stroke patients. The impression is more frequent measurements of blood pressure, serum glucose, troponin and supplementary computer tomography or magnetic resonance imaging.

DETAILED DESCRIPTION:
There is in general a focus on misuse of health resources. An increasing amount of guidelines is produced to reduce the variation in treatment of patients with the same diagnosis. Many recommendations are weak but seems though to have considerable impact on in hospital care. The issues to be studied are all grounded on weak clinical evidence. A pilot study confirmed the suspicion of very frequent measurements of blood pressure, glucose, troponin and frequent supplementary CT and MRI. The intention is to study these issues in a larger population including an evaluation of utility of the different examinations and evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of stroke according to ICD 10th revision (code I61 I63 and I64)
* Hospitalized between January 1 and December 31, 2015

Exclusion Criteria:

* Previous hospitalization with a diagnosis of stroke in 2015.
* Foreigners and patients from other regions of Norway.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients > 18 years, registered with a diagnosis of stroke during 2015 at Innlandet Hospital Trust Lillehammer.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of supplementary computer tomography and magnetic resonance imaging of the brain. | 3 months
  Number
The number of blood sugar measurements | 72 hours after admission to hospital
  Number

SECONDARY OUTCOMES:
Troponin measurement, | 72 hours
  frequency and level of max value
Number of blood pressure measurement | 72 hours
  Number
Transfer to tertiary center | 72 hours
  Number

CONTACTS AND LOCATIONS:
Overall Officials: Ingebjørg Hartz, Study Director — Sykehuset Innlandet HF
Locations (2):
- Norway (2):
  - Innlandet Hospital Trust Lillehammer, Lillehammer
  - Ellen Bøhmer, Lillehammer

IPD SHARING:
Plan to Share IPD: No